CLINICAL TRIAL: NCT00066677
Title: Phase II and Coagulation Study of rhuMAb-VEGF With or Without Docetaxel in Patients With Previously Treated Metastatic Pancreatic Adenocarcinoma
Brief Title: Bevacizumab With or Without Docetaxel in Treating Patients With Previously Treated Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped accordining to early stopping rule for futility
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316454; P30CA006927 (NIH); FCCC-03003
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhuMAB-VEGF (Experimental): bevacizumab 10 mg/kg by intravenous infusion over 30-90 minutes once every 2 weeks until disease progression, unacceptable toxicity or patient preference.
  Interventions: Drug: rhuMAB-VEGF
- rhuMAB-VEGF and Docetaxel (Experimental): rhuMAB-VEGF,bevacizumab: 10 mg/kg by intravenous infusion over 30-90 minutes once every 2 weeks docetaxel, Taxotere: 35 mg/m2 given intravenously over 1 hour on days 1, 8, and 15 of each 28 day cycle. Treatment continued until evidence of disease progression, unacceptable toxicity, or patient preference.
  Interventions: Drug: rhuMAB-VEGF; Drug: docetaxel

INTERVENTIONS:
Drug: rhuMAB-VEGF
Drug: docetaxel
  Arms: rhuMAB-VEGF and Docetaxel

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining bevacizumab with docetaxel may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying bevacizumab and docetaxel to see how well they work compared to bevacizumab alone in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival of patients with previously treated metastatic pancreatic adenocarcinoma treated with bevacizumab with or without docetaxel.
* Determine the objective response rate and overall survival of patients treated with these regimens.
* Determine the incidence of thromboembolic events in patients treated with these regimens.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and docetaxel IV over 1 hour on days 1, 8, and 15.
* Arm II: Patients receive bevacizumab as in arm I. In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 46 patients (23 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Metastatic disease
* Unidimensionally measurable disease outside of the pancreas

  * At least 1 lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Must have received 1, and only 1, prior gemcitabine-containing regimen for metastatic disease unless disease has recurred within 6 months after treatment with neoadjuvant or adjuvant gemcitabine-containing therapy
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL (transfusion allowed)
* No bleeding diathesis or coagulopathy

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST and ALT no greater than 1.5 times ULN
* INR no greater than ULN
* PTT no greater than ULN

Renal

* Creatinine no greater than 2.0 mg/dL
* No clinically significant renal impairment
* Urine protein:creatinine ratio ≥ 1.0

Cardiovascular

* No prior myocardial infarction
* No prior stroke
* No clinically significant cardiovascular disease
* No uncontrolled hypertension (i.e., blood pressure greater than 160/110 mm Hg on medication)
* No unstable angina
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac dysrhythmia requiring medication
* No peripheral vascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history or evidence of CNS disease (e.g, primary brain tumor or seizures not controlled with standard medical therapy)
* No other medical condition that would preclude study participation
* No psychiatric condition that would preclude study participation
* No other prior or concurrent malignancy that would preclude study participation
* No significant traumatic injury within the past 28 days
* No serious, nonhealing wound, ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic granulocyte or platelet growth factors

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* More than 7 days since prior fine needle aspirations or core biopsies
* More than 28 days since prior surgery (except closed biopsy or access port placement)
* More than 28 days since prior open biopsy
* No concurrent surgery

Other

* More than 4 weeks since prior experimental drug study participation
* More than 4 weeks since prior investigational drugs
* No other concurrent experimental drug study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-10; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Cohen, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Astsaturov IA, Meropol NJ, Alpaugh RK, Burtness BA, Cheng JD, McLaughlin S, Rogatko A, Xu Z, Watson JC, Weiner LM, Cohen SJ. Phase II and coagulation cascade biomarker study of bevacizumab with or without docetaxel in patients with previously treated metastatic pancreatic adenocarcinoma. Am J Clin Oncol. 2011 Feb;34(1):70-5. doi: 10.1097/COC.0b013e3181d2734a. PMID 20458210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at Fox Chase Cancer Center between October 2004 and December 20006.
Groups:
- rhuMAB-VEGF: rhuMAB-VEGF :
- rhuMAB-VEGF and Docetaxel: rhuMAB-VEGF :
  docetaxel :
Period: Overall Study
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 10 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: 4 months
Population: The study was stopped according to the early stopping rule for futility. All patients who entered the study have died.
Measure: Median (Full Range); unit: days
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel
Number analyzed (Participants) | 16 | 16
days | 43 [28 to 120] | 48 [28 to 120]

2. Secondary Outcome: Objective Response Rate
Time Frame: 56 days
Measure: Number; unit: participants
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel
Number analyzed (Participants) | 16 | 16
participants | 0 | 0

3. Secondary Outcome: Overall Survival
Time Frame: From date of registration until the date of death, assessed up to 5 years
Population: The study was stopped according to the early stopping rule for futility. None of the patients survived.
Measure: Median (Full Range); unit: days
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel
Number analyzed (Participants) | 16 | 16
days | 165 [28 to 480] | 125 [28 to 480]

4. Secondary Outcome: Number of Participants With Thromboembolic Events
Time Frame: 93 days
Measure: Number; unit: participants
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel
Number analyzed (Participants) | 16 | 16
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | rhuMAB-VEGF | rhuMAB-VEGF and Docetaxel
All-Cause Mortality (participants affected / at risk) | 16/16 | 16/16
Serious Adverse Events (participants affected / at risk) | 13/16 | 15/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rhuMAB-VEGF (N=16) | rhuMAB-VEGF and Docetaxel (N=16)
Anorexia (General disorders) | 10 | 11
Cholangitis (General disorders) | 0 | 2
Dehydration (General disorders) | 3 | 4
diarrhea (General disorders) | 3 | 4
DVT/pulmonary embolism (General disorders) | 2 | 2
Dysgeusia (General disorders) | 0 | 3
Fatigue (General disorders) | 13 | 15
GI Bleeding (Gastrointestinal disorders) | 1 | 2
Hyperkalemia (General disorders) | 1 | 2
Hyperuricemia (General disorders) | 2 | 0
Hypoalbuminemia (General disorders) | 9 | 10
Hypertension (General disorders) | 3 | 1
Injection site reaction (General disorders) | 0 | 2
Nail Changes (General disorders) | 0 | 4
Nausea and vomiting (General disorders) | 7 | 9
Parasthesias (General disorders) | 0 | 4
Perforation (General disorders) | 0 | 1
Peritonitis (General disorders) | 1 | 1
Proteinuria (General disorders) | 6 | 8
Watery eyes (General disorders) | 0 | 6
Anemia (Blood and lymphatic system disorders) | 12 | 15
Leukopenia (Blood and lymphatic system disorders) | 5 | 11
Neutropenia (Blood and lymphatic system disorders) | 4 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
The study was stopped according to the early stopping rule for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No